CLINICAL TRIAL: NCT06852092
Title: Study on Mass Balance of [14C]HSK39297 in Healthy Chinese Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HSK39297-102
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C]HSK39297 (Experimental)
  Interventions: Drug: Carbon-14 labeled HSK39297

INTERVENTIONS:
Drug: Carbon-14 labeled HSK39297 — Dose A

SUMMARY:
To evaluate the absorption, metabolism and excretion in healthy Chinese male subjects after a single oral dose of [14C]HSK39297

DETAILED DESCRIPTION:
1. To quantitatively analyze the total radioactivity in excreta after oral administration of [14C]HHSK39297 in healthy subjects, obtain the data on human radioactivity excretion rate and determine the main excretion pathways
2. To quantitatively analyze the total radioactivity in whole blood and plasma in healthy subjects after oral administration of [14C]HSK39297, to obtain the pharmacokinetics of total radioactivity in plasma and to investigate the distribution of total radioactivity in whole blood and plasma
3. To obtain the radioactive metabolite profile in plasma, urine, and feces after oral administration of [14C]HSK39297 in healthy subjects, to identify the main metabolites and to determine the metabolism and elimination pathways

ELIGIBILITY:
Inclusion Criteria:

1. Chinese healthy male subjects aged between 18 and 45 years old (inclusive, at the time of signing the informed consent form);
2. Body weight ≥ 50 kg and body mass index (BMI) within the range of 19 - 26 kg/m² (inclusive);
3. Capable of comprehending the procedures and methodologies of this study, disposed to strictly adhere to the related requirements of the protocol, and capable of signing the informed consent form.

Exclusion Criteria:

1. Abnormal and clinically significant findings in physical examination, vital signs, laboratory tests (blood routine, biochemistry, coagulation function, urine routine, stool routine + fecal occult blood, thyroid function), ophthalmic examination (slit lamp, intraocular pressure, fundus photography), 12 - lead electrocardiogram [QT interval corrected by Fridericia method (QTcF), 350 - 450 ms (inclusive) for men], X - ray chest film (anterior - posterior and lateral views), abdominal B - ultrasound (liver, gallbladder, pancreas, spleen), urinary system B - ultrasound (kidneys, ureters, bladder, prostate), etc.
2. Positive for hepatitis B surface antigen, hepatitis C virus IgG antibody, human immunodeficiency virus antibody and antigen p24, and Treponema pallidum antibody.
3. Use of prescription drugs, over - the - counter drugs, or health care products, including Chinese patent medicine, within 14 days before the screening period or within 5 half - lives of the drug (whichever is longer).
4. Participated in a clinical trial and received investigational drugs or devices within 3 months before screening.
5. Use of any drugs that inhibit or induce the activity of liver drug - metabolizing enzymes or P - gp inhibitors within 30 days before screening.
6. Dysphagia or any conditions that may affect drug absorption (e.g., gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy).
7. Habitual constipation/diarrhea (feces collection required), history of malabsorption syndrome, or severe GI symptoms within 1 week before screening.
8. History of serious diseases in cardiovascular, digestive, etc. systems or other diseases/physiological conditions interfering with trial results.
9. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, atrioventricular block, QT prolongation syndrome, or having symptoms of QT prolongation syndrome and a family history (indicated by genetic evidence or sudden cardiac death of close relatives at a young age).
10. History of capsular bacterial infection (e.g., Neisseria meningitidis, etc.) within 6 months before screening.
11. History of tuberculosis infection or currently suffering from tuberculosis.
12. Underwent major surgery within 6 months before screening or surgical incision not healed (excluding healed appendicitis and rectal prolapse surgeries).
13. Severely allergic, allergic to trial drugs/excipients, two or more other drugs/foods, or having special diet requirements and unable to follow a unified diet.
14. Having hemorrhoids or perianal diseases with regular/ongoing rectal bleeding, irritable bowel syndrome, or inflammatory bowel disease.
15. Alcoholism or regular drinking (> 14 alcohol units/week) within 6 months before screening, or positive alcohol breath test.
16. Smoking more than 5 cigarettes per day or habitually using nicotine - containing products within 3 months before the screening period and being unable to quit during the trial.
17. Having drug abuse or dependence, with a positive urine drug abuse screening.
18. Habitually drinking grapefruit juice or excessive tea (more than 8 cups a day, 1 cup = 250 mL), or excessive caffeine intake (more than 3 cups of coffee a day, etc.) and being unable to quit during the trial.
19. Long - term exposure to radiation at work, or significant radiation exposure (≥ 2 chest/abd CT or ≥ 3 other X - rays) within 1 year before the trial, or participated in a radiopharmaceutical trial within 1 year.
20. Received a live vaccine within 1 month before screening or planned to during the trial.
21. History of fainting at the sight of needles/blood, difficult blood collection, or intolerance to venipuncture.
22. Fertility plan during the trial and within 1 year after the last dose, or disagreed to take strict contraceptive measures.
23. Blood loss or donation ≥ 400 mL within 3 months before screening, or received a blood transfusion within 1 month.
24. For any reason subject is considered by the investigator to be an unsuitable candidate.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Recovery of total radioactivity in urine and fecal samples | Up to 312 hours post dose
  Mass balance recovery of total radioactivity in urine and fecal samples
Total radioactivity in plasma PK | Up to 312 hours post dose.
  PK parameters of total radioactivity in the plasma; Ratio of total radioactivity concentration in whole blood/plasma at different time points.
Percentage of radioactivity and identification of metabolites in plasma, urine and fecal samples | Up to 312 hours post dose.
  Percentage of prototype drugs and its metabolites in plasma, urine and fecal samples. Identification of the major metabolites

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 312 hours post dose.
  All subjects will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms and ophthalmological assessments

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China